CLINICAL TRIAL: NCT03061032
Title: Open-label Study of Efficacy and Safety of Generic Sofosbuvir/Ledipasvir±Ribavirin in Iranian Patients With Hepatitis C Virus Genotype 1 Infection
Brief Title: Treatment of Hepatitis C Virus Infection With Generic Sofosbuvir/Ledipasvir in Iranian Patients
Acronym: HepCC-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Iran Hepatitis Network (Other)
Collaborators: Baqiyatallah Research Center for Gastroenterology and Liver Diseases (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHN10002
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sofosbuvir/Ledipasvir for 12W (Experimental): Patients without cirrhosis and previous history of treatment will be treated with this regimen.
  Daily fixed dose combination of Sofosbuvir (400mg)/Ledipasvir (90 mg) for 12 weeks.
  Interventions: Drug: Sofosbuvir/Ledipasvir 12W
- Sofosbuvir/Ledipasvir+Ribavirin for 12W (Experimental): Patients with compensated cirrhosis and/or previous history of treatment will be treated with this regimen.
  Daily fixed dose combination of Sofosbuvir (400mg)/Ledipasvir (90 mg) plus Daily Ribavirin (1000-1200 mg) for 12 weeks.
  Interventions: Drug: Sofosbuvir/Ledipasvir plus Ribavirin 12W
- Sofosbuvir/Ledipasvir for 24W (Experimental): Patients with compensated or decompensated cirrhosis and/or previous history of treatment and with contraindication of Ribavirin will be treated with this regimen.
  Daily fixed dose combination of Sofosbuvir (400mg)/Ledipasvir (90 mg) for 24 weeks.
  Interventions: Drug: Sofosbuvir/Ledipasvir 24W
- Sofosbuvir/Ledipasvir+Ribavirin for 24W (Experimental): Patients with decompensated cirrhosis will be treated with this regimen. Daily fixed dose combination of Sofosbuvir (400mg)/Ledipasvir (90 mg) plus Daily Ribavirin (1000-1200 mg) for 24 weeks.
  Interventions: Drug: Sofosbuvir/Ledipasvir plus Ribavirin 24W

INTERVENTIONS:
Drug: Sofosbuvir/Ledipasvir 12W — Daily fixed dose combination of Sofosbuvir (400mg)/Ledipasvir (90 mg) for 12 weeks.
  Arms: Sofosbuvir/Ledipasvir for 12W
Drug: Sofosbuvir/Ledipasvir plus Ribavirin 12W — Daily fixed dose combination of Sofosbuvir (400mg)/Ledipasvir (90 mg) plus Daily Ribavirin (1000-1200 mg) for 12 weeks.
  Arms: Sofosbuvir/Ledipasvir+Ribavirin for 12W
Drug: Sofosbuvir/Ledipasvir 24W — Daily fixed dose combination of Sofosbuvir (400mg)/Ledipasvir (90 mg) for 24 weeks.
  Arms: Sofosbuvir/Ledipasvir for 24W
Drug: Sofosbuvir/Ledipasvir plus Ribavirin 24W — Daily fixed dose combination of Sofosbuvir (400mg)/Ledipasvir (90 mg) plus Daily Ribavirin (1000-1200 mg) for 24 weeks.
  Arms: Sofosbuvir/Ledipasvir+Ribavirin for 24W

SUMMARY:
Hepatitis C virus (HCV) infection with around 0.5% and 2.2% prevalence in Iran and world is one of the public health problems resulting in chronic liver disease, cirrhosis and hepatocellular carcinoma. All cases of chronic HCV infections are candidates of treatment to prevent advanced liver diseases. The previous Pegylated-interferon and Ribavirin therapy was not efficient in all cases and results in numerous number of side-effects. Introduction of direct acting antiviral agents (DAAs) such as Sofosbuvir and Ledipasvir make the eradication of HCV possible however these regimens are not affordable and available in developing countries. The generic DAAs are manufactured in many of these countries such as Iran to provide the treatment with reasonable price.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection
* >18 years old

Exclusion Criteria:

* HIV co-infected
* Liver transplanted
* Receiving drugs with suspected interactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Response | 12 weeks after completion of treatment
  Undetectable HCV RNA 12 weeks after completion of treatment with RT-PCR or TMA with a 15 IU/mL limit of detection

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Moayed Alavian, MD, Study Chair — Iran Hepatitis Network; Heidar Sharafi, PhD, Study Director — Iran Hepatitis Network; Bita Behnava, MD, Principal Investigator — Iran Hepatitis Network; Mohammad Saeid Rezaee-Zavareh, MD, Principal Investigator — Iran Hepatitis Network

IPD SHARING:
Plan to Share IPD: Undecided